CLINICAL TRIAL: NCT01145443
Title: A Multicenter Study of the Effect of Intensive Care Unit Attending Physician Work Schedules on Outcomes Relevant to Society
Brief Title: Multicenter Intensivist Weekend Scheduling Study
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Case Western Reserve University (Other); Ohio State University (Other); Indiana University (Other); University of Toledo Health Science Campus (Other)
Responsible Party: Allan Garland / Associate Professor of Medicine & Community Health Sciences, University of Manitoba Faculty of Medicine
Other Study IDs: IRB-05-00307
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Critical Illness; Burnout, Professional
Keywords: Organizational models; Intensive care units; Physicians; Staffing and scheduling; Burnout, professional; Job satisfaction
MeSH Terms: conditions — Critical Illness; Burnout, Professional

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continuous intensivist staffing model: These are the patients admitted to participating Intensive Care Units during the 3 month phases of the study when a single intensivist was the sole attending physician of record for intervals of 2 weeks (or 1/2 month).
  Interventions: Other: Alternative Intensivist staffing models.
- Discontinuous intensivist staffing model: These are the patients admitted to participating Intensive Care Units during the 3 month phases of the study when, for intervals of 2 weeks (or 1/2 month), there was a single intensivist who was the primary attending of record during Mondays-Fridays, but cross-covering colleagues took over that role during the weekends.
  Interventions: Other: Alternative Intensivist staffing models.

INTERVENTIONS:
Other: Alternative Intensivist staffing models. — During the study period, each participating ICU alternated between two distinct intensivist staffing formats: (i) in the Discontinuous arm of the study, there was a weekend cross-coverage format wherein an intensivist was responsible for care for a two week or half-month block, but colleagues covered the weekends within each block, or (ii) in the Continuous arm of the study, there was an uninterrupted staffing format, wherein a single intensivist was responsible for the entire two week, or half-month, period. In each ICU the study interval was divided into three phases, so that the models alternated twice in each ICU, beginning with either the weekend cross-coverage or the uninterrupted staffing formats, the four hospitals were randomly assigned between these two patterns.

SUMMARY:
The care of critically ill patients in Intensive Care Units (ICUs) is an important part of modern health care systems. However, ICU care suffers from similar problems as the rest of the health care system. Powerful arguments support the concept that most of problems in complex systems, such as ICUs, relates to flaws in institutional systems and processes that hinder the ability of individuals to perform their jobs well. To fix these problems, the defective systems and processes must be redesigned in ways that make it easy for people to do their job well, and hard to make mistakes. Altering the structure of ICU care for the purpose of improving ICU performance is an example of Organizational Systems Engineering, alternatively called Total Quality Management.

Another serious problem in ICU care is that after 2007 there will be a increasing shortage of physicians specializing in the care of the critically ill (Intensivists), with a 35% shortfall by 2030. One contributor to this shortage is that Intensivists retire at a younger age than do physicians in general, and often curtail their care of critically ill patients even before they retire. It is likely that the emotional and physical demands of this career choice leads Intensivists to "burn out" and leave the field prematurely. For these reasons it is important to find ways to make working as an Intensivist more sustainable so that the most experienced practitioners will continue in the field up to a normal retirement age.

The way in which groups of Intensivists organize themselves to provide care in an ICU is highly variable. One potentially important way in which Intensivist staffing differs is in the degree of continuity of care. The more days in a row that the same physician cares for a patient the greater the continuity of care. While it is generally held that a higher continuity of care results in better care and better outcomes for patients, in fact there are no studies addressing this issue. On the other side of the coin however, it seems likely that working many days in a row increases the physical and emotional burdens on the Intensivist, increasing job distress and job burnout over time.

A common pattern of Intensivist staffing, in which continuity of care is reduced, is when the Intensivist who is caring for ICU patients during the weekdays has the weekend off, during which one of his/her partners provides "cross-coverage". While it is reasonable to hypothesize that cross-coverage would lead to inefficient patient care, at the same time it may reduce the burdens on the Intensivists.

This purpose of this study is to investigate the effects of weekend cross-coverage on both ICU patients and on Intensivists. This will be a multicenter study performed in 4 member institutions of the Midwest Critical Care Consortium: The University of Toledo, MetroHealth Medical Center, Ohio State University, and Indiana University. Five adult medical ICUs from the six institutions will participate in this study, with two ICUs from the Ohio State University site.

To answer the research questions, each participating ICU will alternate between two common models of Intensivist staffing. In both models an Intensivist is responsible for ICU care for 14 days. In the Continuous model, a single Intensivist will be responsible for all 14 days. In the Discontinuous model, both weekends during the 14 days will be cross-covered by a colleague. Continuity of care is higher in the Continuous model, which has 2 physician transitions over a 4 week period, while the Discontinuous model has 8 transitions per 4 weeks. Each participating ICU will use one model for 12 weeks, then switch to the other model for 12 weeks, and finally revert back to the first model for the final 12 weeks of this 36 week study. To address problems of historical controls, seasonal differences, and to increase comparability of groups, the participating ICUs have been randomly assigned to begin the study either with the Continuous or Discontinuous model.

Comparisons will be made between the two scheduling models in: (1) patient outcomes, specifically hospital mortality rate, ICU length of stay, and hospital length of stay, and (2) Intensivist outcomes, specifically job distress, job burnout, and the balance between work and home life.

Since there is currently nothing known about whether weekend cross-coverage influences medical care, both models of care are common in ICUs. Thus the investigators expect that the findings of this study will have general relevance. While the patients admitted to the participating ICUs during this study would not be expected to benefit from this investigation, the results derived are expected to enable policy makers to make evidence-based decisions about this important aspect of ICU physician staffing and thus improve the performance and/or cost-effectiveness of ICU care, benefiting future ICU patients, and society.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission contained entirely within the period of a single intensivist staffing format during the study period.

Exclusion Criteria:

* Repeat ICU admissions during the study period
* ICU admissions that overlapped more than one intensivist staffing format during the study period

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the participating Intensive Care Units during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1945 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | Up to 32 weeks
  ICU length of stay, measured in hours

SECONDARY OUTCOMES:
ICU mortality | Up to 32 weeks
  Vital status at the end of each patients' ICU admission
Hospital mortality | Up to 1 year
  Vital status at the end of each patient's hospitalization
Hospital length of stay | Up to 1 year
  Length of stay in the hospital, in hours
Job burnout among Intensivists | 2 weeks
  This is a scale obtained from having the Intensivists complete surveys. It is derived from the National Study of the Changing Workforce, a large, national survey of U.S. workers performed every five years by the Families and Work Institute, and formerly performed for decades by the Unites States Department of Labor.
Job stress among Intensivists | 2 weeks
  This is a scale obtained from having the Intensivists complete surveys. It is derived from the National Study of the Changing Workforce, a large, national survey of U.S. workers performed every five years by the Families and Work Institute, and formerly performed for decades by the Unites States Department of Labor.
Imbalance between work and personal life among Intensivists | 2 weeks
  This is a scale obtained from having the Intensivists complete surveys. It is derived from the National Study of the Changing Workforce, a large, national survey of U.S. workers performed every five years by the Families and Work Institute, and formerly performed for decades by the Unites States Department of Labor.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Indiana University Hospital, Indianapolis, Indiana
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio

REFERENCES:
- [Derived] Ali NA, Hammersley J, Hoffmann SP, O'Brien JM Jr, Phillips GS, Rashkin M, Warren E, Garland A; Midwest Critical Care Consortium. Continuity of care in intensive care units: a cluster-randomized trial of intensivist staffing. Am J Respir Crit Care Med. 2011 Oct 1;184(7):803-8. doi: 10.1164/rccm.201103-0555OC. PMID 21719756